CLINICAL TRIAL: NCT01753557
Title: A Phase 3 Study of MP-424 in Combination With PEG-IFN Alfa-2a and RBV, in Subjects With Genotype 1 Hepatitis C, Who Are Treatment-Naïve or Relapsed After Previous Treatment
Brief Title: Efficacy and Safety of MP-424, Peginterferon Alfa-2a (PEG-IFN Alfa-2a), and Ribavirin(RBV) in Treatment-Naïve or Relapsed Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G060-A12
Record Dates: First submitted 2012-12-13; First posted 2012-12-20 (Estimated); Results first posted 2016-10-03 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Chronic Hepatitis C (CHC)
Keywords: Pegasys
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment-Naive (Experimental)
  Interventions: Drug: MP-424; Drug: RBV; Drug: PEG-IFN alfa-2a
- Treatment-Relapsed (Experimental)
  Interventions: Drug: MP-424; Drug: RBV; Drug: PEG-IFN alfa-2a

INTERVENTIONS:
Drug: MP-424 — MP-424: 750mg every 8 hours (q8h) for 12 weeks
Drug: RBV — RBV: 600 - 1000 mg/day based on body weight for 24 weeks
Drug: PEG-IFN alfa-2a — PEG-IFN alfa-2a: 180mcg/week for 24 weeks

SUMMARY:
This study will evaluate the efficacy and safety of MP-424 with PEG-IFN Alfa-2a and RBV in patients with genotype 1 hepatitis C, who are naïve to its treatment or relapsed after previous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Genotype 1 CHC
* treatment-naïve or relapsers (patient who relapsed after previous treatment)
* Able and willing to follow contraception requirements

Exclusion Criteria:

* Cirrhosis of the liver or hepatic failure
* Hepatitis B surface antigen-positive or HIV (Human Immunodeficiency Virus) antibodies-positive
* History of, or concurrent hepatocellular carcinoma
* History of, or concurrent depression, schizophrenia, or suicide attempt in the past
* Pregnant, lactating, or suspected pregnant patients, or male patients whose female partner is pregnant

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuoki Kondo, M.D., Study Director — Tanabe Pharma Corporation
Locations (1):
- Toranomon Hospital, Kawasaki, Takatsu-ku, Japan

REFERENCES:
- [Result] Kumada H, Suzuki F, Kamiya N, Orihashi M, Nakayasu Y, Yamada I. Efficacy and safety of telaprevir with pegylated interferon alpha-2a and ribavirin in Japanese patients. Hepatol Res. 2017 May;47(6):514-521. doi: 10.1111/hepr.12722. Epub 2016 Jun 4. PMID 27062488

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment-Naive; Treatment-Relapsed: Drug: MP-424 (generic name:Telaprevir) 750mg every 8 hours(q8h) for 12 weeks Drug: RBV (Ribavirin) 600 - 1000 mg/day based on body weight for 24 weeks Drug: PEG-IFN alfa-2a 180mcg/kg/week for 24 weeks
Period: Overall Study
Arm/Group | Treatment-Naive | Treatment-Relapsed
Started | 35 | 19
Completed | 35 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment-Naive; Treatment-Relapsed: Drug: MP-424 750mg q8h for 12 weeks Drug: RBV 600 - 1000 mg/day based on body weight for 24 weeks Drug: PEG-IFN alfa-2a 180mcg/kg/week for 24 weeks
- Total: Total of all reporting groups
Arm/Group | Treatment-Naive | Treatment-Relapsed | Total
Number analyzed (Participants) | 35 | 19 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (10.5) | 54.3 (9.5) | 52.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 26 | 10 | 36

OUTCOME MEASURES:

1. Primary Outcome: Undetectable HCV (Hepatitis C Virus) RNA (Ribonucleic Acid) at 24 Weeks After Completion of Drug Administration (SVR, Sustained Viral Response)
Time Frame: 48 weeks
Measure: Number (95% Confidence Interval); unit: percentage of subjects achieving SVR
Arm/Group | Treatment-Naive | Treatment-Relapsed
Number analyzed (Participants) | 35 | 19
percentage of subjects achieving SVR | 85.7 [69.7 to 95.2] | 94.7 [74.0 to 99.9]

2. Secondary Outcome: Undetectable HCV RNA at 4 Weeks After Beginning of Drug Administration (RVR, Rapid Viral Response)
Time Frame: 4 weeks
Measure: Number (95% Confidence Interval); unit: percentage of subjects achieving RVR
Arm/Group | Treatment-Naive | Treatment-Relapsed
Number analyzed (Participants) | 35 | 19
percentage of subjects achieving RVR | 88.6 [73.3 to 96.8] | 100.0 [82.4 to 100.0]

3. Secondary Outcome: Undetectable HCV RNA at Completion of Drug Administration (ETR, End-of-treatment Response)
Time Frame: 24 weeks
Measure: Number (95% Confidence Interval); unit: percentage of subjects achieving ETR
Arm/Group | Treatment-Naive | Treatment-Relapsed
Number analyzed (Participants) | 35 | 19
percentage of subjects achieving ETR | 97.1 [85.1 to 99.9] | 100.0 [82.4 to 100.0]

4. Secondary Outcome: Undetectable HCV RNA at 12 Weeks After Completion of Drug Administration
Time Frame: 36 weeks
Measure: Number (95% Confidence Interval); unit: percentage of subjects achieving SVR12
Arm/Group | Treatment-Naive | Treatment-Relapsed
Number analyzed (Participants) | 35 | 19
percentage of subjects achieving SVR12 | 82.9 [66.4 to 93.4] | 94.7 [74.0 to 99.9]

5. Secondary Outcome: Transition of Serum HCV RNA Levels
Time Frame: baseline，Day2，Day3，1Weeks，2Weeks，3Weeks，4Weeks，End of treatment，Follow-up 12weeks，Follow-up 24weeks
Measure: Median (Inter-Quartile Range); unit: log IU/mL
Arm/Group | Treatment-Naive | Treatment-Relapsed
Number analyzed (Participants) | 35 | 19
log IU/mL
  baseline (n=35,19) | 6.70 [6.30 to 7.15] | 7.05 [6.30 to 7.30]
  Day2 (n=35,19) | 3.80 [3.60 to 4.20] | 4.00 [3.70 to 4.30]
  Day3 (n=35,19) | 3.10 [3.00 to 3.50] | 3.30 [3.00 to 3.50]
  1Weeks (n=35,19) | 2.00 [1.60 to 2.50] | 2.00 [1.70 to 2.50]
  2Weeks (n=34,19) | 1.00 [0.50 to 1.00] | 1.00 [0.50 to 1.30]
  3Weeks (n=35,19) | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 1.00]
  4Weeks (n=35,19) | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 0.50]
  End of treatment (n=35,19) | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 0.50]
  Follow-up 12Weeks (n=33,19) | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 0.50]
  Follow-up 24Weeks (n=35,19) | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 0.50]

6. Secondary Outcome: Viral Sequencing at the Non-structural 3 Protease Region of HCV Virus（Result of Resistance-associated Variants Analysis)
Time Frame: From baseline to 24 weeks after completion of drug administration
Measure: Number; unit: participants
Groups:
- Treatment-Naïve; Treatment-Relapsed: Drug: MP-424 750mg q8h for 12 weeks Drug: RBV 600 - 1000 mg/day based on body weight for 24 weeks Drug: PEG-IFN alfa-2a 180mcg/kg/week for 24 weeks
Arm/Group | Treatment-Naïve | Treatment-Relapsed
Number analyzed (Participants) | 4 | 1
participants
  V36A | 1 | 0
  T54A | 0 | 1
  Not detected | 3 | 0

ADVERSE EVENTS:
Arm/Group | Treatment-Naive | Treatment-Relapsed
Serious Adverse Events (participants affected / at risk) | 0/35 | 2/19
Other Adverse Events (participants affected / at risk) | 35/35 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-Naive (N=35) | Treatment-Relapsed (N=19)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-Naive (N=35) | Treatment-Relapsed (N=19)
Nasopharyngitis (Infections and infestations) | 14 | 6
Periodontitis (Infections and infestations) | 3 | 2
Anaemia (Blood and lymphatic system disorders) | 33 | 19
Hypothyroidism (Endocrine disorders) | 2 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 7 | 8
Decreased appetite (Metabolism and nutrition disorders) | 6 | 11
Insomnia (Psychiatric disorders) | 6 | 5
Headache (Nervous system disorders) | 15 | 8
Dysgeusia (Nervous system disorders) | 7 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 8 | 3
Nausea (Gastrointestinal disorders) | 7 | 9
Stomatitis (Gastrointestinal disorders) | 5 | 7
Vomiting (Gastrointestinal disorders) | 5 | 3
Abdominal discomfort (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 13 | 6
Drug eruption (Skin and subcutaneous tissue disorders) | 11 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 7
Renal impairment (Renal and urinary disorders) | 3 | 2
Pyrexia (General disorders) | 20 | 10
Malaise (General disorders) | 16 | 12
Injection site erythema (General disorders) | 14 | 3
Injection site reaction (General disorders) | 4 | 4
Thirst (General disorders) | 2 | 2
White blood cell count decreased (Investigations) | 29 | 14
Platelet count decreased (Investigations) | 29 | 13
Blood uric acid increased (Investigations) | 21 | 6
Blood creatinine increased (Investigations) | 18 | 5
Blood bilirubin increased (Investigations) | 8 | 2
Blood triglycerides increased (Investigations) | 6 | 1
Hyaluronic acid increased (Investigations) | 5 | 4
Blood potassium decreased (Investigations) | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Folliculitis (Infections and infestations) | 1 | 1
Hordeolum (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 0 | 3
Oral herpes (Infections and infestations) | 0 | 2
Furuncle (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Enterocolitis viral (Infections and infestations) | 0 | 1
Lipid metabolism disorder (Metabolism and nutrition disorders) | 0 | 1
Depressive symptom (Psychiatric disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Retinopathy (Eye disorders) | 8 | 0
Vision blurred (Eye disorders) | 1 | 1
Asthenopia (Eye disorders) | 2 | 0
Eye pain (Eye disorders) | 2 | 0
Dry eye (Eye disorders) | 1 | 1
Retinal haemorrhage (Eye disorders) | 1 | 1
Cataract (Eye disorders) | 0 | 1
Eye discharge (Eye disorders) | 0 | 1
Punctate keratitis (Eye disorders) | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 4
Hepatic steatosis (Hepatobiliary disorders) | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 1 | 2
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 0
Feeling hot (General disorders) | 1 | 1
Liver function test abnormal (Investigations) | 3 | 0
Neutrophil count decreased (Investigations) | 3 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 1
Blood phosphorus decreased (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Bilirubin conjugated increased (Investigations) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other